CLINICAL TRIAL: NCT03821181
Title: Remote Ischemic Conditioning Prevents Ischemic Cerebrovascular Events In Children With Moyamoya Disease: A Randomized Controlled Trial
Brief Title: The Effect of RIC on TIA/Stroke in Children With Moyamoya Disease
Acronym: RIC-PMD-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Collaborators: 307 Hospital of PLA (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIC-PMD-1
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Moyamoya Disease; TIA; Children; Stroke
Keywords: pediatric moyamoya disease; TIA; Stroke; Remote ischemic conditioning
MeSH Terms: conditions — Moyamoya Disease; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Interventions: Device: RIC group
- sham group (Sham Comparator): patients allocated to the sham group will undergo a sham RIC procedure during which bilateral arm cuffs are inflated to a pressure of 30 mmHg for five cycles of 5 min, followed by 5 min of relaxation of the cuffs.
  Interventions: Device: Sham group

INTERVENTIONS:
Device: RIC group — Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: RIC group
Device: Sham group — patients allocated to the sham group will undergo a sham RIC procedure during which bilateral arm cuffs are inflated to a pressure of 30 mmHg for five cycles of 5 min, followed by 5 min of relaxation of the cuffs.
  Arms: sham group

SUMMARY:
Moyamoya disease is a common reason of transient ischemic attack (TIA) and stroke in children. Remote ischemic conditioning (RIC) has been shown to prevent recurrent stroke in intracranial arterial stenosis, but it is unclear whether RIC can prevent TIA or stroke in children with moyamoya disease. This study aims to evaluate the effect of RIC on TIA/stroke in children with moyamoya disease.

DETAILED DESCRIPTION:
This study will provide insights into the preliminary proof of principle, safety, and efficacy of RIC in pediatric MMD patients, and this data will provide parameters for future larger scale clinical trials if efficacious

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥0 and ≤18
* all of the patients underwent digital subtraction angiography and met the current diagnostic criteria recommended by the Research Committee on MMD (Spontaneous Occlusion of the Circle of Willis) of the Ministry of Health and Welfare of Japan in 2012
* The CVR of patients detected by SPECT is not impaired severely
* The patients didn't suffer stroke before.
* Informed consent obtained from patient or acceptable patient's surrogate

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Severe hemostatic disorder or severe coagulation dysfunction
* Patients with unilateral MMD or the presence of secondary moyamoya phenomenon caused by autoimmune disease, Down syndrome, neurofibromatosis, leptospiral infection, or previous skull-base radiation therapy
* Any of the following cardiac disease - rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with participation
* Serious, advanced, or terminal illnesses with anticipated life expectancy of less than one year
* Patient participating in a study involving other drug or device trial study
* Patients with existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Unlikely to be available for follow-up for 3 months
* Contraindication for RIC - severe soft-tissue injury, fracture, or peripheral vascular disease in the upper limbs.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of transient ischemic attack(TIA) | during baseline to 12months after therapy
  TIA means transient ischemic attack, two neurologists will evaluate patients with ischemic symptoms and make diagnosis.magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
The incidence rate of ischemic stroke | during baseline to 12months after therapy
  Two neurologists will evaluate patients with ischemic symptoms and make diagnosis.magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.

SECONDARY OUTCOMES:
Cerebral perfusion | change from baseline to 12months after therapy
  cerebral perfusion status in the operation side at 12 months posttreatment as assessed by single photon emission computed tomography (SPECT).
The mean blood flow velocity of cerebral vascular detected by TCCD | changes form baseline to 6months，12months after therapy
  TCCD means tran-scranial color-coded duplex sonography.
The score of National Institute of Health stroke scale score | during baseline to 12months after therapy
  National Institute of Health Stroke Scale (NIHSS) is considered as a standardized assessment of neurological functions in the acute phase of stroke, and it is generally used to quantify patient's neurological impairments on 15 items in 11 fields of different neurological status.The score of the scale ranges from 0 to 42.And higher score indicates worse neurological function.The NHISS will be assessed by certified study investigator, who is blinded to the treatment assignment.
The score of Modified Rankin scale score | during baseline to 12months after therapy
  The Modified Rankin Scale Score (mRS) is the most comprehensive and most widely used primary outcome measurement to assess the neurological functional disability in contemporary acute stroke trials. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranges from 0 (no symptom) to 5 (severe disability) and 6 (death). The investigators will use mRS to evaluate the degree of disability or dependence during daily activities. The mRS will be assessed by certified study investigator, who is blinded to the treatment assignment.
Incidence rate of symptomatic intracerebral hemorrhage | during baseline to 12months after therapy
  Symptomatic intracranial hemorrhage, including any subarachnoid hemorrhage associated with clinical symptoms and symptomatic intracerebral hemorrhage. Head computed tomography or magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
The number of cerebral lacunar infarction | changes from baseline to 12months after therapy
  magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
The volume of cerebral lacunar infarction | changes from baseline to 12 months after therapy
  magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
The rate of death and adverse event | during baseline to 12months after therapy
  All causes of death will be included to compute mortality at 12 months after therapy
Number of distal radial pulses | changes from baseline to 6, 12months after therapy
  professional doctors will check the distal radial pulses
Visual inspection of local edema of fundus oculi | changes from baseline to 6, 12months after therapy
  Professional oculists will visually inspect the fundus oculi to evaluate whether there is local edema.
The number of patients with erythema,and/or skin lesions related to RIC | changes from baseline to 6, 12months after therapy
  Professional doctors will check it and the investigator will record the number.
Palpation for tenderness | changes from baseline to 6, 12months after therapy
  Professional doctors will definite whether there's a palpation for tenderness
The number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | during baseline to 12months after therapy
  The investigator will record the number.
The number of patients with any other adverse events related to RIC intervention | during baseline to 12months after therapy
  The investigator will record the number.
The score of ABCD2 | during baseline to 12months after therapy
  When subjects are diagnosed as TIA within 12 months after therapy ,The investigators use this scale to evaluate the patients' risk of stroke who with TIA .The score of the scale ranges from 0 to 7, and the higher score indicates higher risk of stroke in the patients who with TIA.The scale will be assessed by qualified investigator who are blinded to the treatment assignment.
The level of S-100A4 | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of matrix metalloproteinase 9 (MMP-9) | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of basic fibroblast growth factor | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of platelet derived growth factor | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of vascular endothelial growth factor | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of hs-CRP(high-sensitive C-reactive protein) | change from baseline (pre-RIC treatment) to 6 months ,12 months after therapy
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
cerebral perfusion examined by SPECT | from baseline（pre-RIC treatment) to 12 months after therapy
  cerebral perfusion status post-treatment will be assessed by single photon emission computed tomography (SPECT).
cerebral perfusion examined by ASL | from baseline（pre-RIC treatment) to 12 months after therapy
  cerebral perfusion status post-treatment will be assessed by arterial spin labeling(ASL)
variant of the RNF-213 gene | from baseline（pre-RIC treatment) to 12 months after therapy
  The investigators will save the blood sample in -20℃，and detect the variant RNF-213 gene

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China